CLINICAL TRIAL: NCT02242461
Title: Rhodiola Crenulata as an Adjunctive Therapy in Patients With Chronic Obstructive Pulmonary Disease
Brief Title: Rhodiola Crenulata as an Adjunctive Therapy in COPD
Acronym: COPD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Chung Shan Medical University (Other)
Responsible Party: Principal Investigator, GCRC, Chief, Department of Critical Care Medicine and Division of Pulmonary Medicine, Chung Shan Medical University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CS11144
Record Dates: First submitted 2014-09-04; First posted 2014-09-17 (Estimated); Last update posted 2014-09-17 (Estimated); Status verified 2014-09

CONDITIONS: COPD
Keywords: COPD, Rhodiola L., clinical trial, biomarkers, spirometry
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Rhodiola placebo capsules (Placebo Comparator): starch
  Interventions: Drug: Rhodiola placebo capsules
- Rhodiola Crenulata (Experimental): Rhodiola Crenulata
  Interventions: Drug: Rhodiola Crenulata

INTERVENTIONS:
Drug: Rhodiola placebo capsules — Corn starch
  Arms: Rhodiola placebo capsules
Drug: Rhodiola Crenulata — Rhodiola Crenulata
  Other Names: Rhodiola
  Arms: Rhodiola Crenulata

SUMMARY:
We hypothesize that add-on Rhodiola L extract capsule to the regimen of patients with moderate-to-severe COPD (1) may provide a potential of systemic effects of anti-inflammation and anti-oxidation for these patients, and these effects (2) may reflect in the improvement of patients' physiological measurements, quality of life and exercise tolerance.

DETAILED DESCRIPTION:
This is a single center, randomized, double-blind, placebo controlled clinical trial.

Eligibility criteria:

1. moderate-to-severe COPD patients
2. aged 40-80 years,
3. abstaining from cigarette smoking or maintaining a stable dose of cigarette consumption,
4. no acute exacerbation of COPD,
5. clinically being stable for one month and longer,
6. not undergoing exercise training program.

Primary endpoint:

six-minute walk distance in meters at week 12.

ELIGIBILITY:
Inclusion Criteria:

1. moderate-to-severe COPD patients
2. aged 40-80 years,
3. abstaining from cigarette smoking or maintaining a stable dose of cigarette consumption,
4. no acute exacerbation of COPD,
5. clinically being stable for one month and longer,
6. not undergoing exercise training program.

Exclusion Criteria:

1. uncontrolled diabetes mellitus by plasma fasting sugar >200 mg/dl,
2. uremia or CKD stage 5,
3. chronic heart failureby NYFC III,
4. cerebrovascular disease,
5. uncontrolled anemia by Hb < 10 mg/dl,
6. active malignant diseases,
7. other hospitalized acute illness,
8. systemic prednisolone > 10 mg per day.

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2012-05; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
six-minute walk distance in meters at week 12. | 12 weeks

SECONDARY OUTCOMES:
mid-arm circumference and triceps skin thickness, Borg scale, COPD assessment test score, St. George Respiratory disease questionnaire, hospital anxiety and depression scale(HADS) and maximum cardiopulmonary exercise test | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Ming Lung Chuang, Principal Investigator — Department of Critical Care Medicine and Division of Pulmonary Medicine
Locations (1):
- Department of Critical Care Medicine and Division of Pulmonary Medicine, Dawan, Ming-Lung Chuang, Taiwan

REFERENCES:
- [Derived] Chuang ML, Wu TC, Wang YT, Wang YC, Tsao TC, Wei JC, Chen CY, Lin IF. Adjunctive Treatment with Rhodiola Crenulata in Patients with Chronic Obstructive Pulmonary Disease--A Randomized Placebo Controlled Double Blind Clinical Trial. PLoS One. 2015 Jun 22;10(6):e0128142. doi: 10.1371/journal.pone.0128142. eCollection 2015. PMID 26098419